CLINICAL TRIAL: NCT04051905
Title: Evolution of Bone Volume in the Mandibular Posterior Area After Natural Healing and Flapless Technique
Brief Title: Bone Loss in Posterior Mandible Postextraction Sockets
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0395
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Guided Bone
Keywords: Regeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the bone loss after extraction. The surgery protocol is flapless, and the teeth are mandibular premolars or molars leaving sockets with 4 walls intact or at least 3 walls intact and the buccal wall at 80% . This study will include 40 patients

DETAILED DESCRIPTION:
Primary objective :

Estimate the percentage of bone volume loss o and the percentage thickness loss of the buccal and palatal cortical for patients who underwent natural healing in the mandibular molar and premolar areas.

Methods :

Before tooth extraction of a premolar or molar in mandibular area by flapless technique, a CBCT preoperative is performed to verify the integrity of cortical and measure the height and width of the residual cavity. Caliper measurements will also be performed during surgery in order to integrate also the thickness of the bone tables and gingival thickness.

After natural healing , the pre-implant scan performed at six months postoperatively will measure the height and width of the grafted cell, to compare measurements and evaluate the dynamics of alveolar resorption.

ELIGIBILITY:
Inclusion criteria

* patients requiring tooth extraction
* aged 18 to 80
* Patients showing no indication against-General to surgery

Exclusion criteria

* Patient with against-indication for surgical treatment.
* Patients with an important loss of vestibular cortical
* Patients requiring and accepting a bone graft
* Unstabilized periodontal disease or aesthetic indication.
* Inability to maintain a good level of oral hygiene and good cooperation.
* Higher tobacco consumption has 10cig / day
* Acute dental infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of patients aged between 18 and 80 years with one to two posterior mandibular teeth to extract in absence of bone graft and able to benefit from a flapless technique.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Cone beam diagnostic examination | Day diagnostic (Day 0)
  Cone beam diagnostic examination: Millimeter measurements will be taken at Day 0.
  This examination is an X-ray technique that uses a cone-shaped radiation beam. The measurements will be made on radiographic examinations
  Mucous measures
  * Vestibular cortical Distance, lingual cortical measured in the middle of the cell
  * Depth of the slot lingual cortical side
  * Depth of the cell vestibular cortical side
  Bone measures
  * Thickness of the lingual cortical measured caliper 2 millimeters under the rim
  * Vestibular cortical thickness measured with calipers 2 millimeters under the rim
  * Depth of the slot lingual cortical side
  * Depth of the cell vestibular cortical side

SECONDARY OUTCOMES:
Cone beam pre implant examination | 5 or 6 months
  Cone beam pre implant examination : millimeter measurements will be taken at 5 or 6 months.
  This examination is an X-ray technique that uses a cone-shaped radiation beam. The measurements will be made on radiographic examinations
  Mucous measures
  * Vestibular cortical Distance, lingual cortical measured in the middle of the cell
  * Depth of the slot lingual cortical side
  * Depth of the cell vestibular cortical side
  Bone measures
  * Thickness of the lingual cortical measured caliper 2 millimeters under the rim
  * Vestibular cortical thickness measured with calipers 2 millimeters under the rim
  * Depth of the slot lingual cortical side
  * Depth of the cell vestibular cortical side
Clinical measures | Day of surgery
  Clinical measures on the day of surgery
  Bone measures
  * Thickness of the lingual cortical measured caliper 2 millimeters under the rim
  * Vestibular cortical thickness measured with calipers 2 millimeters under the rim
  * Cortical vestibular cortical lingual distance, measured in the middle of the cell
  * Depth of the slot lingual cortical side
  * Depth of the cell vestibular cortical side
  Mucous measure:
  * Gum buccal keratinized
  * Keratinized gingiva lingual
  * Cortical vestibular cortical lingual distance measured in the middle of the cell

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BOUSQUET, MCU PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UHMontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC